CLINICAL TRIAL: NCT05769647
Title: Effect of Two Different Methods Applied During Peripheral Intravenous Catheter Placement on Pain and Anxiety
Brief Title: Effect of Two Different Methods on Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serpil SU, Assistant Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nec EU
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-12

CONDITIONS: Pain
Keywords: Peripheral Intravenous Catheter Insertion; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients will be informed about the study and their consent will be obtained without explaining which group they are in. Since the researcher manages the implementation process of the study, researcher blinding cannot be done. In addition, it will be ensured that the researcher learns which group the patients are in after the patients accept to participate in the study. Thus, the internal validity of the research will be ensured. Since data is collected from the patients in the sample group at the time of admission to the ward, interaction between patients will be prevented.
  At the same time, blind technique will be applied in terms of statistical analysis in the research. The data will be recorded on the computer by the researcher without using the expression of experimental and control groups, and data analysis will be done by another statistician other than the person who made the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Glasses Group (Experimental): * "Volunteer Information and Approval Form" will be filled.
  * Physician request, the name and surname of the individual will be checked.
  * Patient Information Form and State Anxiety Scale will be filled.
  * The video containing the nature walk will be watched by virtual reality. 3 minutes after the individual starts watching the video, the IV catheter insertion attempt will be performed while continuing to watch the video.
  * Visual Pain Scale and State Anxiety Scale will be filled within one minute after intravenous catheter placement is completed.
  Interventions: Device: Virtual Reality Glasses
- Ball Squeezing Group (Experimental): * "Volunteer Information and Approval Form" will be filled.
  * Physician request, the name and surname of the individual will be checked.
  * Patient Information Form and State Anxiety Scale will be filled.
  * Patients will be given a ball and instructed to tighten and loosen with their free hand during IVC placement. The IV catheter insertion attempt will be made while the patient continues to squeeze the ball.
  * Visual Pain Scale and State Anxiety Scale will be filled within one minute after intravenous catheter placement is completed.
  Interventions: Device: Stress Ball
- Control Group: (No Intervention): * "Volunteer Information and Approval Form" will be filled.
  * Physician request, the name and surname of the individual will be checked.
  * Patient Information Form and State Anxiety Scale will be filled.
  * An intravenous catheter will be placed.
  * Visual Pain Scale and State Anxiety Scale will be filled within one minute after intravenous catheter placement is completed.

INTERVENTIONS:
Device: Virtual Reality Glasses — 3 minutes after the individual starts watching the video, the IV catheter insertion attempt will be performed while continuing to watch the video.
  Arms: Virtual Reality Glasses Group
Device: Stress Ball — Patients will be given a ball and instructed to tighten and loosen with their free hand during IVC placement. The patient will continue to squeeze the ball throughout the IV catheter insertion attempt.
  Arms: Ball Squeezing Group

SUMMARY:
The aim of this study is to determine the effect of virtual reality glasses and ball squeezing method used during peripheral intravenous catheter placement on pain and anxiety.The hypotheses of this research are that virtual reality glasses and a stress ball reduces pain and anxiety.

DETAILED DESCRIPTION:
This study was designed as a pretest-posttest regular parallel group, randomized controlled experimental. The research will be carried out in the general surgery clinic of Necmettin Erbakan University Meram Medical Faculty Hospital. Patients will be randomly assigned to three groups: ball squeezing (37), virtual reality glasses (37) and control group (37). For Virtual Reality Glasses Group: The video containing the nature walk will be watched by virtual reality. 3 minutes after the individual starts watching the video, the IV catheter insertion attempt will be performed while continuing to watch the video. For Ball Squeezing Group: Patients will be given a ball and instructed to tighten and loosen with their free hand during intravenöz catheter placement. The intravenöz catheter insertion attempt will be made while the patient continues to squeeze the ball. For Control Group: No application will be made during intravenous catheter placement in the control group.The primary outcome of this study was to determine the patients' pain scores during the peripheral venous cannula insertion process.The secondary outcomes of the study were to determine the patients' anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the General Surgery clinic.
* No verbal, perceptual and visual communication problems,
* Being between 18 - 65 years old,
* Being literate,
* Volunteer to participate in the research,
* Not using drugs that will create a chronic analgesic effect,
* Absence of chronic or acute pain,
* No intervention in the last month in the vein where an IV catheter was placed.
* The absence of scar tissue and infection in the areas to be used for IV catheter placement,
* It was determined as not having a disease (such as neuropathy) that would cause problems in feeling pain.

Exclusion Criteria:

* The individual's desire to leave the study,
* Inability to perform the ball squeezing motion,
* Feeling unwell during IV catheter placement (such as dizziness, palpitations),
* During use of VR, the patient experiences symptoms such as nausea and dizziness,
* Using sedatives or alcohol,

Termination criteria

• Failure of PIV catheter placement,

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Pain evaluated using the Visual Pain Scale | It will be applied within 1 minute after the virtual reality reality glasses and ball squeezing processes.
  The Visual Pain Scale is mostly a 10 cm/100 mm long horizontal or vertical line starting with "No pain" and ending with "Unbearable pain". While measuring, there is no pain at one end, very severe or unbearable pain is written on the other end, and the patient marks his or her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.

SECONDARY OUTCOMES:
Anxiety evaluated using the State Anxiety Scale | It will be applied before and afte within 1 minute after the virtual reality reality glasses and ball squeezing processes.
  In the State Anxiety Inventory, the individual evaluates how he or she feels "at the moment" and according to the severity of the emotions or behaviors expressed in the items (1) "never", (2) "a little", (3) "a lot" and (4) "a lot". are asked to choose one of the statements "completely". The highest score of 4 is given for choosing the phrase "completely", and the lowest score is 1 for choosing the phrase "not at all". The lowest total score that can be obtained from the State Anxiety Scale is 20, and the highest total score is 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil SU, Principal Investigator — Necmettin Erbakan University
Locations (2):
- Turkey (Türkiye) (2):
  - Necmettin Erbakan University, Konya
  - Turkey, Necmettin Erbakan University, Konya

IPD SHARING:
Plan to Share IPD: No